CLINICAL TRIAL: NCT04147247
Title: An Open-label, Phase I Trial to Determine the Maximum-tolerated Dose and Investigate Safety, Pharmacokinetics and Efficacy of BI 905681 Administered Intravenously in Patients With Advanced Solid Tumours
Brief Title: A Trial to Find the Safe Dose for BI 905681 in Patients With Incurable Tumours or Tumours That Have Spread
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1424-0001; 2019-003490-25 (EudraCT Number)
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 1.0 milligram/kilogram BI 905681 (Experimental): Subjects received an intravenous infusion of 1.0 milligram/kilogram BI 905681 on day 1 of each cycle (1 cycle = 21 days). Patients may continue on treatment for unlimited cycles, until criteria for stopping treatment are met.
  Interventions: Drug: BI 905681
- 2.5 milligram/kilogram BI 905681 (Experimental): Subjects received an intravenous infusion of 2.5 milligram/kilogram BI 905681 on day 1 of each cycle (1 cycle = 21 days). Patients may continue on treatment for unlimited cycles, until criteria for stopping treatment are met.
  Interventions: Drug: BI 905681
- 5.0 milligram/kilogram BI 905681 (Experimental): Subjects received an intravenous infusion of 5.0 milligram/kilogram BI 905681 on day 1 of each cycle (1 cycle = 21 days). Patients may continue on treatment for unlimited cycles, until criteria for stopping treatment are met.
  Interventions: Drug: BI 905681
- 7.0 milligram/kilogram BI 905681 (Experimental): Subjects received an intravenous infusion of 7.0 milligram/kilogram BI 905681 on day 1 of each cycle (1 cycle = 21 days). Patients may continue on treatment for unlimited cycles, until criteria for stopping treatment are met.
  Interventions: Drug: BI 905681
- 8.5 milligram/kilogram BI 905681 (Experimental): Subjects received an intravenous infusion of 8.5 milligram/kilogram BI 905681 on day 1 of each cycle (1 cycle = 21 days). Patients may continue on treatment for unlimited cycles, until criteria for stopping treatment are met.
  Interventions: Drug: BI 905681

INTERVENTIONS:
Drug: BI 905681 — Infusion

SUMMARY:
The primary objective of this trial is to determine the maximum tolerated dose (MTD)/optimal biological dose (OBD) of BI 905681 given as an intravenous infusion and to determine the recommended dose and dosing schedule for further trials in the development of BI 905681. The MTD will be defined based on the frequency of patients experiencing dose-limiting toxicities (DLTs) during the MTD/DLT evaluation period, which is defined as the first cycle of treatment. Separate MTDs will be determined for Schedule A and Schedule B.

The secondary objective of the trial is to determine the pharmacokinetic (PK) profile of BI 905681.

DETAILED DESCRIPTION:
Study was opened to recruitment until 29-Oct-2021, however from 15-Apr-2021 no patient was recruited.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of an advanced, unresectable and/or metastatic non-haematologic malignancy. Patient must have measurable or evaluable lesions (according to Response Evaluation Criteria in Solid Tumours (RECIST) v 1.1).
* Patient who has failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options.
* Patients willing to undergo mandatory tumour biopsy at the time points specified in the protocol.
* Eastern Cooperative Oncology Group (ECOG) Score of 0 or 1 (R01-0787).
* Adequate organ function defined as all of the following:

  * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L; haemoglobin ≥9.0 g/dL; platelets ≥100 x 10^9/L without the use of haematopoietic growth factors within 4 weeks of start of study medication.
  * Total bilirubin ≤1.5 x the upper limit of normal (ULN), except for patients with Gilbert's syndrome: total bilirubin ≤3 x ULN or direct bilirubin ≤1.5 x ULN.
  * Creatinine ≤1.5 x ULN. If creatinine is >1.5 x ULN, patient is eligible if concurrent creatinine clearance ≥50 ml/min (measured or calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula or Japanese version of CKD-EPI formula for Japanese patients).
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 x ULN if no demonstrable liver metastases, or otherwise ≤5 x ULN
  * Alkaline Phosphatase (ALP) <5 x ULN
* At least 18 years of age at the time of consent or over the legal age of consent in countries where that is greater than 18 years.
* Signed and dated written informed consent in accordance with International Conference on Harmonisation (ICH) - Good Clinical Practice (GCP) and local legislation prior to admission to the trial
* Life expectancy ≥3 months at the start of treatment in the opinion of the investigator
* Further inclusion criteria apply

Exclusion criteria:

* Osteoporosis ≥ CTCAE Grade 2
* Osteoporotic compression fracture within 12 months prior to informed consent which is clinically significant in the opinion of the investigator.
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase I, open-label, non-randomised dose-escalation study of BI 905681 administered intravenously as a single agent in patients with advanced solid tumors.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | 1.0 Milligram/Kilogram BI 905681 | 2.5 Milligram/Kilogram BI 905681 | 5.0 Milligram/Kilogram BI 905681 | 7.0 Milligram/Kilogram BI 905681 | 8.5 Milligram/Kilogram BI 905681
Started | 3 | 4 | 5 | 4 | 5
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 5 | 4 | 5
Not completed — Progressive disease | 3 | 3 | 4 | 4 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Clinical Disease Progression | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): includes all patients who received at least one infusion of BI 905681.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.0 Milligram/Kilogram BI 905681 | 2.5 Milligram/Kilogram BI 905681 | 5.0 Milligram/Kilogram BI 905681 | 7.0 Milligram/Kilogram BI 905681 | 8.5 Milligram/Kilogram BI 905681 | Total
Number analyzed (Participants) | 3 | 4 | 5 | 4 | 5 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (6.5) | 63.8 (2.1) | 55.6 (17.6) | 66.3 (11.1) | 62.0 (9.6) | 60.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 1 | 2 | 10
  Male | 0 | 3 | 2 | 3 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 4 | 4 | 5 | 19
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 1 | 4
  White | 3 | 2 | 1 | 4 | 4 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD)/Optimal Biological Dose (OBD) of BI 905681
Description: The MTD/OBD of BI 905681. The MTD will be assessed based on the number of patients experiencing Dose Limiting Toxicities (DLTs), graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, in the first cycle of treatment (3 weeks). The MTD is defined as the highest dose with less than 25% risk of the true DLT rate being equal to or above 33%.
Time Frame: The first cycle of treatment, up to 21 days.
Population: MTD Evaluation Set (MTDS): includes all patients who received at least one infusion of BI 905681 and who were not replaced for the MTD determination.
Measure: Number; unit: milligram/kilogram
Groups:
- BI 905681: Comprises all dose cohorts during the dose escalation phase. Subjects received an intravenous infusion of BI 905681 on day 1 of each cycle (1 cycle = 21 days).
Arm/Group | BI 905681
Number analyzed (Participants) | 18
milligram/kilogram | NA — The MTD could not be determined due to the prematurely discontinuation of the trial. The trial was completed according to protocol but stopped early due to a lack of response.

2. Primary Outcome: Number of Patients Experiencing Adverse Events (AEs) During the Entire Treatment Period
Description: Number of patients experiencing adverse events (AEs) during the entire treatment period.
Time Frame: From the first administration of study till the last administration of study drug +42 days, up to 126 days.
Population: Treated Set (TS): includes all patients who received at least one infusion of BI 905681.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.0 Milligram/Kilogram BI 905681 | 2.5 Milligram/Kilogram BI 905681 | 5.0 Milligram/Kilogram BI 905681 | 7.0 Milligram/Kilogram BI 905681 | 8.5 Milligram/Kilogram BI 905681
Number analyzed (Participants) | 3 | 4 | 5 | 4 | 5
Participants | 2 | 4 | 5 | 4 | 4

3. Secondary Outcome: Cmax: Maximum Measured Concentration of BI 905681 in Serum After First Infusion
Description: Cmax: maximum measured concentration of BI 905681 in serum after first infusion.
Time Frame: 5 minutes before and 1, 1.5, 4, 8, 24, 72, 168, 336 and 504 (5 minutes before 2nd infusion) hours following the first infusion.
Population: Pharmacokinetics Analysis Set (PKS): All patients who received at least one infusion of BI 905681 and who provide at least one observation for at least one pharmacokinetic (PK) endpoint without important protocol violations relevant to the evaluation of PK. two subjects were excluded, one subject due to having a prolonged infusion (1mg/kg group) and one subject (8.5 mg/kg group) was not able to receive the full dose due to safety reasons.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | 1.0 Milligram/Kilogram BI 905681 | 2.5 Milligram/Kilogram BI 905681 | 5.0 Milligram/Kilogram BI 905681 | 7.0 Milligram/Kilogram BI 905681 | 8.5 Milligram/Kilogram BI 905681
Number analyzed (Participants) | 2 | 4 | 5 | 4 | 4
microgram/milliliter | NA (NA) — not calculable with two subjects. | 49.6 (19.7) | 157 (18.0) | 185 (23.1) | 201 (21.4)

4. Secondary Outcome: AUC0-tz: Area Under the Serum Concentration-time Curve Over the Time Interval From 0 to the Last Measured Time Point (tz)
Description: AUC0-tz: area under the serum concentration-time curve over the time interval from 0 to the last measured time point (tz).
Time Frame: as for outcome 3
Population: Pharmacokinetics Analysis Set (PKS): All patients who received at least one infusion of BI 905681 and who provide at least one observation for at least one pharmacokinetic (PK) endpoint without important protocol violations relevant to the evaluation of PK. one subject (8.5 mg/kg group) was excluded due to not being able to receive the full dose for safety reasons.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter
Arm/Group | 1.0 Milligram/Kilogram BI 905681 | 2.5 Milligram/Kilogram BI 905681 | 5.0 Milligram/Kilogram BI 905681 | 7.0 Milligram/Kilogram BI 905681 | 8.5 Milligram/Kilogram BI 905681
Number analyzed (Participants) | 3 | 4 | 5 | 4 | 4
hour*microgram/milliliter | 4260 (27.8) | 7640 (10.6) | 18200 (53.2) | 30000 (23.8) | 18900 (217)

ADVERSE EVENTS:
Time Frame: From the first administration of study till the last administration of study drug +42 to 49 days, up to 133 days.
Description: Treated Set (TS): includes all patients who received at least one infusion of BI 905681.
Arm/Group | 1.0 Milligram/Kilogram BI 905681 | 2.5 Milligram/Kilogram BI 905681 | 5.0 Milligram/Kilogram BI 905681 | 7.0 Milligram/Kilogram BI 905681 | 8.5 Milligram/Kilogram BI 905681
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 2/5 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 2/5 | 1/4 | 0/5
Other Adverse Events (participants affected / at risk) | 2/3 | 4/4 | 5/5 | 4/4 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.0 Milligram/Kilogram BI 905681 (N=3) | 2.5 Milligram/Kilogram BI 905681 (N=4) | 5.0 Milligram/Kilogram BI 905681 (N=5) | 7.0 Milligram/Kilogram BI 905681 (N=4) | 8.5 Milligram/Kilogram BI 905681 (N=5)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1.0 Milligram/Kilogram BI 905681 (N=3) | 2.5 Milligram/Kilogram BI 905681 (N=4) | 5.0 Milligram/Kilogram BI 905681 (N=5) | 7.0 Milligram/Kilogram BI 905681 (N=4) | 8.5 Milligram/Kilogram BI 905681 (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 3
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
C-telopeptide increased (Investigations) | 0 | 0 | 1 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Trial was prematurely discontinued due to limited antitumor activity (i.e., lack of a single objective response) & difficulty in enrolling patients with RNF43 (Ring Finger Protein 43) mutations or R-spondin fusions who were willing to undergo a biopsy. The trial aimed to test two schedules for BI 905681 (A: every three weeks in a 3-week cycle, B: every 2 weeks in a 4-week cycle). Maximum tolerated dose/Recommended Phase 2 dose for Schedule A could not be determined, schedule B was not pursued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04147247/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT04147247/SAP_001.pdf